CLINICAL TRIAL: NCT04903457
Title: Investigation of Compensational Mechanism and Effect of Transcranial Direct Stimulation on Motor Learning Through Neural Network Analysis in Stroke Patients
Brief Title: The Effect of tDCS on Motor Learning and Neural Network in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, Principal Investigator, Samsung Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-04-075
Record Dates: First submitted 2021-05-23; First posted 2021-05-26 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real stimulation before motor learning training (Experimental): Patients receive five sessions of tDCS stimulation over C3 (patient with left-sided lesion) or C4 (patient with right-sided lesion) based on 10-20 system immediately before sequential finger tapping task.
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Motor learning
- Sham stimulation before motor learning training (Active Comparator): Patients receive five sessions of sham stimulation over C3 (patient with left-sided lesion) or C4 (patient with right-sided lesion) based on 10-20 system immediately before sequential finger tapping task.
  Interventions: Behavioral: Motor learning

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial direct current stimulation is a form of noninvasive neuromodulation that uses constant and low direct current delivered via electrodes on the scalp.
  Arms: Real stimulation before motor learning training
Behavioral: Motor learning — Sequential finger tapping task training is applied to stroke patients.

SUMMARY:
This study is to investigate the effect of transcranial direct current stimulation (tDCS) simulation on motor learning to stroke patients compared to sham stimulation

ELIGIBILITY:
Inclusion Criteria:

* Unilateral stroke including basal ganglia lesion patients
* Chronic patients over 6 months after onset
* Patients with the movement of fingers

Exclusion Criteria:

* History of psychiatric disease
* Significant other neurological diseases except for stroke
* Difficult to perform this experiment
* Patients who are deemed difficult to participate in this research by the investigator
* Patients with metal implants and medical devices
* History of epilepsy
* Pregnancy
* Skin defect at the site of electrode attachment

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | Baseline, immediately after five brain stimulation sessions
  The score is a stroke-specific, performance-based impairment index. The degree of impairment of upper and lower limbs is measured.

SECONDARY OUTCOMES:
Changes in cortical activity using fNIRS signals during brain stimulation | Baseline, during, immediately after five brain stimulation sessions
  Cortical activities before, during and after brain stimulation sessions are compared.
Changes in motor evoked potential | Baseline, immediately after five brain stimulation sessions
  Resting motor threshold (rMT) and amplitude of motor evoked potential in first dorsal interosseous muscle are measured. These outcomes are measured by transcranial magnetic stimulation over the motor hotspot. The rMT is defined as the minimum stimulus intensity that produced a minimal motor evoked response at rest. The amplitude means peak to peak of the muscle response.
9-hole pegboard test | Baseline, immediately after five brain stimulation sessions
  The test is a standardized, quantitative assessment used to measure finger dexterity of a patient.
Grip & Tip pinch strength test | Baseline, immediately after five brain stimulation sessions
  The test is to measure the maximum isometric strength of hand, forearm, and finger muscles.
Box & Block test | Baseline, immediately after five brain stimulation sessions
  The test is used to measure the gross manual dexterity of a patient, or of a person using an upper limb prosthetic device.
Sequential Finger tapping test | Baseline, immediately after five brain stimulation sessions
  Response time is measured during sequential finger tapping task.
Jebsen-Taylor hand function test | Baseline, immediately after five brain stimulation sessions
  This test is a standardized and objective measure of fine and gross motor hand function using simulated activities of daily living (ADL).

OTHER OUTCOMES:
Resting-state functional MRI | Baseline (Before stimulation sessions)
  Before intervention, MRI is acquired to extract brain characteristics of stroke patients.
Changes in cortical activity using fNIRS signals. | Baseline (Before stimulation sessions)
  Before intervention, fNIRS image is acquired to extract cortical activation of stroke patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea